CLINICAL TRIAL: NCT02221479
Title: A Randomized, Open-label, Two-arm Parallel Group, Comparative Study for Assessing the Clinical Benefit of Subcutaneous Injection of Plerixafor Plus G-CSF for Mobilization and Collection of Peripheral Hematopoietic Stem Cells in Japanese Patients With Multiple Myeloma
Brief Title: Plerixafor Plus Granulocyte Colony-stimulating Factor (G-CSF) For Mobilization And Collection Of Peripheral Hematopoietic Stem Cells In Japanese Participants With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACT13710; U1111-1152-4403 (Other: UTN)
Record Dates: First submitted 2014-08-19; First posted 2014-08-20 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-08

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — plerixafor; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Granulocyte colony-stimulating factor (G-CSF) alone (Active Comparator): G-CSF administered up to 8 days
  Interventions: Drug: Filgrastim
- G-CSF plus plerixafor (Experimental): G-CSF administered up to 8 days (Day 1 to Day 8) and plerixafor administered for 4 days (Day 4 to Day 7)
  Interventions: Drug: plerixafor GZ316455; Drug: Filgrastim

INTERVENTIONS:
Drug: plerixafor GZ316455 — Pharmaceutical form:vial Route of administration: subcutaneous injection
  Other Names: Mozobil
  Arms: G-CSF plus plerixafor
Drug: Filgrastim — Pharmaceutical form:vial Route of administration: subcutaneous injection

SUMMARY:
Primary Objective:

To determine if Multi Myeloma (MM) patients mobilized with granulocyte colony-stimulating factor (G-CSF) plus plerixafor 240 μg/kg are more likely to achieve a target number of greater than or equal to 6 x 10^6 cluster of differentiation (CD) 34+ cells/kg in 2 or fewer days of apheresis than MM patients mobilized with G-CSF alone.

Secondary Objectives:

* To evaluate the safety of G-CSF plus plerixafor arm compared to G-CSF arm in MM patients.
* To compare the 2 treatment arms with respect to the number of participants who achieved a minimum of 2 x 10^6 CD34+ cells/kg in 4 or fewer days of apheresis.
* To compare the 2 treatment arms with respect to the number of days of apheresis required to reach the target of greater than or equal to 6 x 10^6 CD34+ cells/kg.

DETAILED DESCRIPTION:
Total study duration for a participant can be approximately up to 68 days.

ELIGIBILITY:
Inclusion criteria:

* Age 20 to 75.
* Japanese participants with histological or pathological diagnosis of MM.
* First or second complete response (CR) or partial response (PR).

Exclusion criteria:

* Leukemia participants.
* Myelodysplastic syndrome (MDS) participants.
* Less than 2 weeks since completion of last cycle of chemotherapy.
* Failed previous hematopoietic stem cell (HSC) collections or collection attempts.
* Prior autologous or allogeneic transplant.
* Diagnosis of another malignancy.
* Known hypersensitivity to plerixafor, G-CSF or their components.
* Bone marrow involvement greater than 10%.
* Eastern Cooperative Oncology Group (ECOG) performance status greater than 1.
* Not yet recovered from all acute toxic effects of prior Chemotherapy.
* White blood cell (WBC) count less than or equal to 2.5 × 10^9 cells/L.
* Absolute neutrophil count (ANC) less than or equal to 1.5 × 10^9 cells /L.
* Platelet count less than or equal to 100 × 10^9 cells /L.
* Creatinine clearance less than 50 mL/min.
* Aspartate aminotransferase (AST), or alanine aminotransferase (ALT) greater than or equal to 2.5 x upper limit of normal,Total Bilirubin greater than or equal to 2.5 x upper limit of normal.
* Cardiac and pulmonary status insufficient to undergo apheresis or transplantation.
* Active central nervous system (CNS) involvement, active brain metastases, or any history of carcinomatous meningitis.
* Active infection, including unexplained fever (greater than 38 degrees C), or antibiotic therapy within 7 days prior to the first dose of GCSF.
* Less than 6 weeks off nitrosoureas prior to first dose of G-CSF.
* Conditions/situations such as: received prior radio-immunotherapy with ibritumomab tiuxetan or tositumomab iodine, and received radiation therapy to the pelvis.
* Significant concomitant illness, including psychiatric condition that, in the opinion of the Investigator or Sponsor, would adversely affect the participant's participation in the study.
* Abnormal electrocardiogram (ECG) with clinically significant rhythm disturbance (ventricular arrhythmias) or other conduction abnormality in the last year that, in the opinion of the Investigator(s), warrants exclusion of the participants from the trial.
* Previously received experimental therapy within 4 weeks of randomization or who are currently enrolled in another experimental protocol during the G-CSF and plerixafor treatment period.
* Any malignancy related to immunodeficiency virus (HIV) or solid organ transplant; history of known HIV, unresolved viral hepatitis as documented at the detection of hepatitis B surface antigen (HBsAg), hepatitis B surface antibody (HBsAb)[exclude patients who clearly received vaccination], hepatitis B core antibody (HBcAb), and/or hepatitis C virus (HCV) antibody at the time of the screening visit.
* Unwillingness and inability to comply with scheduled visits, drug administration plan, laboratory tests, other study procedures, and study restrictions.
* Related to the active comparator and/or mandatory background therapies.
* Received G-CSF within 7 days prior to the first dose of G-CSF for mobilization.
* Related to the current knowledge of Sanofi compound.
* Pregnant or breast-feeding women.
* All participants, who are sexually active (males and females), must agree to an effective method of contraception while on study treatment and for at least 3 months following plerixafor treatment (including both female participants of child-bearing potential and male participants with partners of childbearing potential).
* Patient who has withdrawn consent before enrollment/randomization.
* Despite screening of the patient, enrollment/randomization is stopped at the study level.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who achieve a collection of greater than or equal to 6 x10^6 cells/kg CD34+ cells in less than or equal to 2 days of apheresis | Day 5 to Day 8 of the apheresis/treatment period

SECONDARY OUTCOMES:
Proportion of participants who achieve a collection of a minimum target of 2 x10^6 cells/kg CD34+ cells in less than or equal to 4 days of apheresis | Day 5 to Day 8 of the apheresis/treatment period
Number of days of apheresis to collect 6 x10^6 cells/kg CD34+ cells | Day 5 to Day 8 of the apheresis/treatment period
Number of days of apheresis to collect 2 x10^6 cells/kg CD34+ cells | Day 5 to Day 8 of the apheresis/treatment period
Total number of CD34+ cells/kg collected over up to 4 apheresis | Day 5 to Day 8 of the apheresis/treatment period
The relative increase (ratio) of peripheral blood CD34+ cell count (cells/μL) | From Day 4 morning to Day 5 morning for both arms, from Day 4 morning to Day 4 evening for GP arm only, and from Day 4 evening to Day 5 morning for GP arm only
Number of participants with adverse events | Up to 68 days
Change from baseline in clinical laboratory measurements | Up to 68 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (5):
- Japan (5):
  - Investigational Site Number 392105, Kamogawa-Shi
  - Investigational Site Number 392103, Kyoto
  - Investigational Site Number 392102, Nagoya
  - Investigational Site Number 392104, Okayama
  - Investigational Site Number 392101, Shibuya-Ku